CLINICAL TRIAL: NCT06977607
Title: Comparative Study Between Platelet- Rich Fibrin Versus Nano-Fat in Improving Facial Nerve Regeneration After Traumatic Injury
Brief Title: Neurorrhaphy Only vs Neurorrhaphy Plus PRF vs Neurorrhaphy Plus Nano-fat in Management of Traumatic Facial Nerve Injury
Acronym: facialinjury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mohie Selim, Specialist, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRF vs Nanofat in VII injury
Record Dates: First submitted 2025-01-16; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Facial Nerve Injuries; Facial Trauma
Keywords: PRF; nanofat; facial nerve
MeSH Terms: conditions — Facial Nerve Injuries

STUDY DESIGN:
Intervention Model Description: * Twenty-one Patients will be randomly assigned to Groups A, B, or C ( 3 equal groups).
  * A research Nurse will perform simple randomization before surgery using the closed-envelop technique.
  * Twenty-one closed envelopes will be used; each 7 carries one of the three groups that will be randomly withdrawn at the time of surgery.
Masking Description: Sample Size and Group Allocation: A total of 21 patients will be randomly assigned to one of three groups: A, B, or C, with 7 patients in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelets Rich Fibrin (Experimental): Injection of PRF, which contains various growth factors, including GDNF and nerve growth factor (NGF), promotes peripheral nerve regeneration post-neurorrhaphy.
  To compare the outcome of Neurorrhaphy Platelet-rich fibrin versus Neurorrhaphy alone and Neurorrhaphy with Nanofat.
  Interventions: Procedure: Platelets Rich Fibrin
- Repair only (Experimental): Neurorrhaphy is the traditional method of surgical repair To compare the outcome of Neurorrhaphy alone Versus Using Different Adjuvants with Neurorrhaphy, such as Platelet-Rich Fibrin and Nano-fat.
  Interventions: Procedure: Repair only
- Nano-fat stem cells (NFSCs) (Experimental): Injection of NFSCs contains abundant stromal vascular fraction cells and adipose-derived stem cells that help tissue regeneration. Post-neurorrhaphy injection contains abundant stromal cells that support tissue regeneration.
  To compare the outcome of Neurorrhaphy with Nanofat-derived stem cells injection versus Neurorrhaphy with platelet-rich fibrin injection.
  Interventions: Procedure: Nano-fat stem cells (NFSCs)

INTERVENTIONS:
Procedure: Platelets Rich Fibrin — Repair of facial nerve injury plus Platelets Rich Fibrin will be injected around the repair and measure the out come in comparison with (Repair only) and (Repair Plus Nano-fat stem cells)
  Other Names: PRF
  Arms: Platelets Rich Fibrin
Procedure: Nano-fat stem cells (NFSCs) — Repair of facial nerve injury plus Nano fat derived stem cells will be injected around the repair and measure the out come in comparison with (Repair only) and (Repair Plus Platelets Rich Fibrin).
  Other Names: NFSCs
  Arms: Nano-fat stem cells (NFSCs)
Procedure: Repair only — facial nerve neurorrhaphy only (repair only) after acute facial nerve trauma and measure the out come in comparison with (Repair plus Nano- fat Stem Cells) and (Repair Plus Platelets Rich Fibrin).
  Other Names: facial nerve neurorrhaphy
  Arms: Repair only

SUMMARY:
The current clinical trial aims to identify the most significant intervention that improves the outcome of post-traumatic facial nerve injury by comparing the following different modalities: neurorrhaphy alone, neurorrhaphy with PRF injection, and neurorrhaphy with Nanofat stem cells graft injection for significantly better Facial nerve regeneration.

DETAILED DESCRIPTION:
Despite advances in microsurgical technology and an improved understanding of nerve regeneration, obtaining satisfactory results after facial nerve injury remains a challenging clinical problem.

Traumatic facial nerve injury may account for up to 10% of the causes of facial nerve palsy and has devastating effects on patients both functionally, emotionally, and aesthetically.

The most common traumatic causes of facial paralysis are resection of tumors, temporal bone fractures, and penetrating trauma to the facial nerve, including iatrogenic injury.

Patients with Facial paralysis are at a higher risk of developing adverse psychological outcomes such as depression, anxiety, and disrupted social interaction.

Facial paralysis has implications for patients' quality of life due to the facial nerve's role in myriad activities of daily living.

Peripheral nerve injuries can result in significant morbidity, including motor and/or sensory loss, which can significantly affect the life of the patient. Nowadays, the gold standard for treating nerve sections is end-to-end neurorrhaphy. Unlike other tissues in the body, peripheral nerve regeneration is slow and usually incomplete. Despite current surgical techniques, less than half of the patients who undergo nerve repair after injury regain good to excellent motor or sensory function. Primary neurorrhaphy is the preferred reconstruction modality over nerve grafting, especially for motor nerves. The main limitation to primary repair is often dictated by tension secondary to increased nerve defect length.

If coaptation without tension is impossible, a cable graft interposition using the greater auricular or sural nerves may be necessary. The success rate of nerve repair, defined as a return to House-Brackmann grade III function or better, varies from 5% to 86% within the literature.

Several new neural repair technologies have been developed recently, such as nerve regeneration bridging technology, electrical stimulation technology, and stem cell therapy technology.

Nanofat is a relatively novel technique in fat grafting that has gained significant interest in regenerative medicine, aesthetics, and translational research. It involves the extraction of autologous fat from a patient, which is then transformed into "nanofat", consisting of small fat particles with a diameter of less than 0.1 mm and containing high concentrations of stem cells and growth factors.

Adipose-derived stem cells have a huge proliferative capacity and can differentiate into mesoderm, ectoderm, and endoderm lineages. Using nano-fat graft, a better quality and faster rate of new epithelium formation in the donor site is possible.

The use of platelets for regenerative medicine has increased in recent years. Platelets, which contain growth factors, play significant roles in cell migration, proliferation, differentiation, and angiogenesis and are associated with the tissue regeneration process.

The use of PRP has increased exponentially in tissue regeneration due to its high therapeutic potential in regenerative medicine. It has been shown that the concentration of platelets compared to basal levels improves the regenerative capacity of cells, tissues, and organs.

Platelet-rich concentrates are used as a source of growth factors to improve the healing process. The diverse preparation protocols and the gaps in knowledge of their biological properties complicate the interpretation of clinical results.

The centrifugation of venous blood produces autologous platelet concentrates (APCs) at different speeds, along with the use or non-use of thrombin and anticoagulants. The fibrin clot formed after this process contains platelets and leukocytes. There are several generations of APCs.

The use of stem cells is a medical biotechnology breakthrough, bringing regenerative therapy into a new era. Stem cells are effective therapeutic agents against several diseases due to their tissue protective and repair mechanisms.

The purpose of this clinical trial is to apply potential therapeutic methods for facial nerve regeneration for acute traumatic facial nerve injury Grade V according to Sunderland classification and compare the outcome of neurorrhaphy, a surgical technique for nerve repair, versus neurorrhaphy plus PRF versus neurorrhaphy plus NFSCs in improving traumatic facial nerve injuries.

ELIGIBILITY:
Inclusion Criteria:

* Recent Facial nerve injury within the first 24 hours of trauma.
* Grade V according to Sunderland classification.

Exclusion Criteria:

* Diabetes Mellitus.
* Steroid Dependent.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Physical examination of the affected facial muscles after injury and Record the time taken for the first muscle excursion to occur following each facial nerve repair modality | 12 months
  **Record the First Occurrence of Muscle Excursion and Movement by facial nerve Physical examination**
  Based on monthly follow-up records Physical examination of the facial muscles affected after the nerve repair is done.
  Record the time taken for the first muscle excursion ( movement) to occur following each facial nerve repair modality.
  Comparing the time interval for each modality - the earlier the occurrence, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M. Selim, Specialist, Principal Investigator — University of Assiut
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
International publishing after finishing the study and the results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: two years
Access Criteria: open access
URL: https://www.aun.edu.eg/main/

REFERENCES:
- [Background] Mijiritsky E, Assaf HD, Peleg O, Shacham M, Cerroni L, Mangani L. Use of PRP, PRF and CGF in Periodontal Regeneration and Facial Rejuvenation-A Narrative Review. Biology (Basel). 2021 Apr 10;10(4):317. doi: 10.3390/biology10040317. PMID 33920204
- [Background] Cecerska-Heryc E, Goszka M, Serwin N, Roszak M, Grygorcewicz B, Heryc R, Dolegowska B. Applications of the regenerative capacity of platelets in modern medicine. Cytokine Growth Factor Rev. 2022 Apr;64:84-94. doi: 10.1016/j.cytogfr.2021.11.003. Epub 2021 Dec 2. PMID 34924312
- [Background] ElSherbeny K, Elshahat A, Gad A. Effect of Nano Fat Graft on the Healing of Donor Site of Split Thickness Skin Graft. The Egyptian Journal of Plastic and Reconstructive Surgery. 2023 Apr 1;47(2):79-88.
- [Background] La Padula S, Ponzo M, Lombardi M, Iazzetta V, Errico C, Polverino G, Russo F, D'Andrea L, Hersant B, Meningaud JP, Salzano G, Pensato R. Nanofat in Plastic Reconstructive, Regenerative, and Aesthetic Surgery: A Review of Advancements in Face-Focused Applications. J Clin Med. 2023 Jun 28;12(13):4351. doi: 10.3390/jcm12134351. PMID 37445386
- [Background] Zou X, Dong Y, Alhaskawi A, Zhou H, Ezzi SHA, Kota VG, Abdulla MHAH, Abdalbary SA, Lu H, Wang C. Techniques and graft materials for repairing peripheral nerve defects. Front Neurol. 2024 Jan 22;14:1307883. doi: 10.3389/fneur.2023.1307883. eCollection 2023. PMID 38318237
- [Background] Gray KM, Burkat AJ, Arney LA, Peterman NJ, Mandala SR, Capito AE. Timing and Predictors of Upper Extremity Peripheral Nerve Reconstruction. JPRAS Open. 2025 Feb 27;44:308-315. doi: 10.1016/j.jpra.2025.02.018. eCollection 2025 Jun. PMID 40271482
- [Background] Grinsell D, Keating CP. Peripheral nerve reconstruction after injury: a review of clinical and experimental therapies. Biomed Res Int. 2014;2014:698256. doi: 10.1155/2014/698256. Epub 2014 Sep 3. PMID 25276813
- [Background] Bassilios Habre S, Bond G, Jing XL, Kostopoulos E, Wallace RD, Konofaos P. The Surgical Management of Nerve Gaps: Present and Future. Ann Plast Surg. 2018 Mar;80(3):252-261. doi: 10.1097/SAP.0000000000001252. PMID 29166306
- [Background] Sasaki R, Watanabe Y, Yamato M, Okamoto T. Tissue-engineered nerve guides with mesenchymal stem cells in the facial nerve regeneration. Neurochem Int. 2021 Sep;148:105062. doi: 10.1016/j.neuint.2021.105062. Epub 2021 May 15. PMID 34004239
- [Background] Vargo M, Ding P, Sacco M, Duggal R, Genther DJ, Ciolek PJ, Byrne PJ. The psychological and psychosocial effects of facial paralysis: A review. J Plast Reconstr Aesthet Surg. 2023 Aug;83:423-430. doi: 10.1016/j.bjps.2023.05.027. Epub 2023 May 19. PMID 37311285
- [Background] Hohman MH, Bhama PK, Hadlock TA. Epidemiology of iatrogenic facial nerve injury: a decade of experience. Laryngoscope. 2014 Jan;124(1):260-5. doi: 10.1002/lary.24117. Epub 2013 Apr 18. PMID 23606475
- [Background] Datta N, Fung E, Hatala A, Melnyk B, Bradley E. Imaging traumatic facial nerve injuries: a narrative review of current strategies and future directions for cranial nerve imaging. Plast Aesthet Res. 2023;10:51. http://dx.doi.org/10.20517/2347-9264.2023.22
- [Background] Yoo MC, Chon J, Jung J, Kim SS, Bae S, Kim SH, Yeo SG. Potential Therapeutic Strategies and Substances for Facial Nerve Regeneration Based on Preclinical Studies. Int J Mol Sci. 2021 May 6;22(9):4926. doi: 10.3390/ijms22094926. PMID 34066483